CLINICAL TRIAL: NCT06352398
Title: Comparison of Analgesic Efficacy in Video-Assisted Thoracoscopic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burcu Bozdogan Tuysuz (Other)
Responsible Party: Sponsor-Investigator, Burcu Bozdogan Tuysuz, Principal Investigator, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBTuysuz
Record Dates: First submitted 2023-12-21; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Video-Assisted Thoracoscopic Surgery
Keywords: Erector spina plan block, postoperative analgesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spina plan block (ESPB) (Active Comparator): erector spina plan block (ESPB) : After providing asepsis and antisepsis conditions to the ESPB group in the sitting position, a high frequency linear USG probe will be placed approximately 2-3 cm lateral to the T5 spinous process in the longitudinal plane. After visualising the T5 transverse process with the in plane approach, the skin will be entered in the craniocaudal direction. Trapezius, rhomboid and erector spinae muscles will be passed and 5 ml of saline will be injected between the erector spinae muscle fascia and vertebral transverse process when the needle rests on the spinous process (approximately 3 cm deep) and the block site will be confirmed. Before the operation 30 ml of 0.25% bupivacaine (1mg/kg) will be injected by negative aspiration.
  Interventions: Procedure: erector spina plan block; Drug: 0.25% bupivacaine
- Serratus posterior superior intercostal plan block (SPSIPB) (Active Comparator): In the SPSIPB group, the patient will be positioned in the lateral position, with the surgical side up and the upper extremity hanging over the patient's head for the USG-guided serratus posterior superior plan block. After asepsis and antisepsis conditions are provided, the spina scapula will be visualised above the scapula with our high frequency linear USG probe. The 3rd rib will be visualised with a high frequency probe medial to the scapula corresponding to the 3rd rib level. The ribs, pleura and the serratus muscle covering it will be determined and the needle tip will be advanced until it touches the 3rd rib.After the 3rd rib is visualised by USG, 5 ml isotonic is given and hydrodissection is performed, 30 ml 0.25% bupivacaine (1mg/kg) will be injected between the serratus posterior superior muscle and the 3rd rib.
  Interventions: Procedure: Serratus posterior superior intercostal plan block (SPSIPB); Drug: 0.25% bupivacaine

INTERVENTIONS:
Procedure: erector spina plan block — erector spina plan block
  Arms: erector spina plan block (ESPB)
Procedure: Serratus posterior superior intercostal plan block (SPSIPB) — Serratus posterior superior intercostal plan block (SPSIPB)
  Arms: Serratus posterior superior intercostal plan block (SPSIPB)
Drug: 0.25% bupivacaine — Before the operation, 0.25% bupivacaine 30 ml was administered to both groups.

SUMMARY:
The 52 patients included in the study were divided into two groups as ESPB (n=26) and SPSIPB (n=26). Before the operation, 0.25% bupivacaine 30 ml was administered to both groups. After admission to the operating room, all patients underwent standard anaesthesia procedures. Morphine 0.05 mg/kg i.v. and parol 1 g i.v. were administered 30 min before the end of the operation. Post operatively the patient was followed up with controlled analgesia. Demographic data, ASA scores, body mass indexes, peri-operative haemodynamic values, remifentanil consumption and duration of surgery were recorded. Post-operative first 24 hours NRS scores, morphine consumption, number of nausea and vomiting episodes were recorded.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of erector spina plan block (ESPB) and Serratus posterior superior intercostal plan block (SPSIPB) on postoperative analgesia management.

After providing asepsis and antisepsis conditions to the ESPB group in the sitting position, a high frequency linear USG probe will be placed approximately 2-3 cm lateral to the T5 spinous process in the longitudinal plane. After visualising the T5 transverse process with the in plane approach, the skin will be entered in the craniocaudal direction. Trapezius, rhomboid and erector spinae muscles will be passed and 5 ml of saline will be injected between the erector spinae muscle fascia and vertebral transverse process when the needle rests on the spinous process (approximately 3 cm deep) and the block site will be confirmed. Then 30 ml of 0.25% bupivacaine (1mg/kg) will be injected by negative aspiration.

In the SPSIPB group, the patient will be positioned in the lateral position, with the surgical side up and the upper extremity hanging over the patient's head for the USG-guided serratus posterior superior plan block. After asepsis and antisepsis conditions are provided, the spina scapula will be visualised above the scapula with our high frequency linear USG probe. The 3rd rib will be visualised with a high frequency probe medial to the scapula corresponding to the 3rd rib level. The ribs, pleura and the serratus muscle covering it will be determined and the needle tip will be advanced until it touches the 3rd rib.After the 3rd rib is visualised by USG, 5 ml isotonic is given and hydrodissection is performed, 30 ml 0.25% bupivacaine (1mg/kg) will be injected between the serratus posterior superior muscle and the 3rd rib. The craniocaudal spread of local anaesthetic will be visualised by USG. Afterwards, the patients will be taken to the operation room and routine monitoring including ECG, peripheral oxygen saturation, non-invasive blood pressure arterial pressure monitoring and bispectral index (BIS) monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 52 healthy volunteers with VATS
* ASA 1-2-3
* 18 to 80 years old

Exclusion Criteria:

* patients with coagulopathy
* wound and infection in the block area
* allergy to local anaesthetic drugs
* mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
morphine consumption first 24 hours | up to 24 hours
  mg

SECONDARY OUTCOMES:
NRS pain score | up to 24 hours
  0 painless to 10 very painful

CONTACTS AND LOCATIONS:
Overall Officials: burcu bozdogan tuysuz, Study Director — medenıyet unıversıty
Locations (1):
- Istanbul Medenıyet Unıversıty, Istanbul, Kadıkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- See also: http — https://pubmed.ncbi.nlm.nih.gov/36883093/